CLINICAL TRIAL: NCT03296969
Title: The Value of Rectus Muscle Re-approximation at Cesarean Delivery
Brief Title: Rectus Muscle Re-approximation at Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Post Cesarean Section Pain
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rectus muscle approximation (Active Comparator): All women underwent Pfnannenstiel incision under general or spinal anaesthesia, with a combination of sharp and blunt dissection to open the abdomen. The rectus muscles are dissected off the fascia, and the muscles are separated in the midline by pulling. Then the uterus is opened followed by fetal and placental extraction. The transverse lower uterine segment incision is closed in two layers of continuous Vicryl number 1 suture. The parietal peritoneum is closed using a continuous absorbable suture. In group (A): rectus muscle re-approximation is done by 3 interrupted sutures, but muscle is not closed in the other group. The rectus sheath is sutured using continuous absorbable sutures. Finally, skin is sutured with subcuticular sutures with Vicryl Rapide
  Interventions: Procedure: cesarean section; Procedure: Rectus muscle approximation
- rectus muscle non approximation (Active Comparator): All women underwent Pfnannenstiel incision under general or spinal anaesthesia, with a combination of sharp and blunt dissection to open the abdomen. The rectus muscles are dissected off the fascia, and the muscles are separated in the midline by pulling. Then the uterus is opened followed by fetal and placental extraction. The transverse lower uterine segment incision is closed in two layers of continuous Vicryl number 1 suture. The parietal peritoneum is closed using a continuous absorbable suture. In group (A): rectus muscle re-approximation is done by 3 interrupted sutures, but muscle is not closed in the other group. The rectus sheath is sutured using continuous absorbable sutures. Finally, skin is sutured with subcuticular sutures with Vicryl Rapide
  Interventions: Procedure: cesarean section

INTERVENTIONS:
Procedure: cesarean section — All women underwent Pfnannenstiel incision under general or spinal anaesthesia, with a combination of sharp and blunt dissection to open the abdomen. The rectus muscles are dissected off the fascia, and the muscles are separated in the midline by pulling. Then the uterus is opened followed by fetal and placental extraction. The transverse lower uterine segment incision is closed in two layers of continuous Vicryl number 1 suture. The parietal peritoneum is closed using a continuous absorbable suture. In group (A): rectus muscle re-approximation is done by 3 interrupted sutures, but muscle is not closed in the other group. The rectus sheath is sutured using continuous absorbable sutures. Finally, skin is sutured with subcuticular sutures with Vicryl Rapide
Procedure: Rectus muscle approximation — aprroximation of the lower parts of rectus abdomius muscles during cesarean section
  Arms: rectus muscle approximation

SUMMARY:
We include in our study 200 pregnant women, primigravidas, at term who underwent elective lower segment Cesarean section for the first time among the age group of 20 - 35 years.

The patients are divided randomly into two groups as follows:

* Group (A): undergoing rectus muscle re-approximation
* Group (B): not undergoing rectus muscle re-approximation

DETAILED DESCRIPTION:
We include in our study 200 pregnant women, primigravidas, at term who underwent elective lower segment Cesarean section for the first time among the age group of 20 - 35 years.

The patients are divided randomly into two groups as follows:

* Group (A): undergoing rectus muscle re-approximation
* Group (B): not undergoing rectus muscle re-approximation
* Examination for diastasis recti abdominis is done for all included patients before delivery, at 6 weeks, and 6 months postpartum. The women are tested in a standardized supine position with arms crossed over the chest. They are instructed to perform an abdominal crunch till the shoulder blades are off the bench. Then we measure the inter-recti distance. If there is no separation or separation ˂ 2 finger breadths so, there is no diastasis recti abdominis. But if the separation is more than 2 finger breadths or more than 4.5 cm so, this is considered diastasis recti abdominis.

The same surgical techniques are used for both groups. All women underwent Pfnannenstiel incision under general or spinal anaesthesia, with a combination of sharp and blunt dissection to open the abdomen. The rectus muscles are dissected off the fascia, and the muscles are separated in the midline by pulling. Then the uterus is opened followed by fetal and placental extraction. The transverse lower uterine segment incision is closed in two layers of continuous Vicryl number 1 suture. The parietal peritoneum is closed using a continuous absorbable suture. In group (A): rectus muscle re-approximation is done by 3 interrupted sutures, but muscle is not closed in the other group. The rectus sheath is sutured using continuous absorbable sutures. Finally, skin is sutured with subcuticular sutures with Vicryl Rapide.

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* undergoing elective Cesarean section

Exclusion Criteria:

* Patients with history of any pelvic or abdominal surgery those having any medical disorder with pregnancy patients with BMI ≥ 40 chronic analgesia use multiple pregnancies

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 4 hours after operation
  • Post-operative pain is analyzed by using 4 point verbal rating scale (VRS) which consists of a list of adjectives describing different levels of pain intensity i.e (no pain =1, mild pain = 2, moderate pain = 3, severe pain = 4), patients are asked to read this list of adjectives and select the word that best describes their level of pain on the scale